CLINICAL TRIAL: NCT01596400
Title: An Open-label, Cross-over, Pharmacokinetic Study to Assess the Safety and Pharmacokinetics of Transdermal Granisetron (Sancuso® Patch) and IV Granisetron in a Pediatric Oncology Population (Aged 13 to 17 Years)
Brief Title: Safety and Pharmacokinetics of Sancuso and IV Granisetron in Patients Aged 13 to 17 Years
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Pharmaceutical Development Ltd (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 392MD/44/C
Record Dates: First submitted 2012-04-26; First posted 2012-05-11 (Estimated); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Chemotherapy Induced Nausea and Vomiting
Keywords: CINV
MeSH Terms: conditions — Vomiting | interventions — Granisetron

ARMS (2):
- Sancuso Arm (Experimental)
  Interventions: Drug: granisetron transdermal system
- IV Granisetron Arm (Active Comparator): IV
  Interventions: Drug: Granisetron IV

INTERVENTIONS:
Drug: granisetron transdermal system — patch
  Other Names: Sancuso
  Arms: Sancuso Arm
Drug: Granisetron IV — IV
  Arms: IV Granisetron Arm

SUMMARY:
The purpose of this study is to determine the dosing strategy for adolescents aged 13 to 17 years.

ELIGIBILITY:
Inclusion Criteria:

1. 13 to 17 years of age inclusive at screening.
2. Written patient or parental (or appropriate legal representative) IRB approved informed consent as appropriate.
3. Written patient assent (as appropriate).
4. Confirmed malignancy.
5. Scheduled to receive 2 or more cycles* of emetogenic chemotherapy requiring 5-HT3 antagonist treatment.
6. Scheduled to receive one or more consecutive days of 5-HT3 antagonist treatment, per cycle, as CINV prophylaxis.

   * The cycles of chemotherapy must be consecutive (i.e. one followed by the other) but do not have to be the first and second cycle of a line of treatment.

Exclusion Criteria:

1. Hypersensitivities, allergies or contraindications to study medications; intolerance of medical tape or sticking plaster.
2. Clinical or laboratory signs and symptoms of significant cerebral, cardiovascular, respiratory, renal, hepatobiliary, pancreatic or infectious disease, which in the Investigator's judgment may interfere with the study assessment or completion of the study.
3. Patients with a known history or predisposition to cardiac conduction interval abnormalities, including QT Syndrome, or known family history of long QT Syndrome or taking medications that are known to prolong the QT interval.
4. Patients scheduled to have routine surgery during the study duration.
5. Patients with a life expectancy of < 6 months.
6. Scarring or significant skin disease on both upper arms.
7. Female patients who are pregnant or breast-feeding. All post menarche female patients must have a pregnancy test at screening.
8. Patients who are known or thought to be sexually active must use effective birth control.**
9. Administration of other investigational drugs within 30 days preceding the screening visit, except for anticancer treatments.
10. Any conditions associated with non-compliance.

    * Effective birth control includes absolute abstinence, or double barrier birth control methods, i.e. condom and one of the following: combined oral contraceptive, diaphragm, depot contraceptive injection.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2012-05; Primary Completion 2015-08 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Plasma concentration | Up to 7 days
  Analysis of the plasma concentration of Intravenous granisetron vs transdermal granisetron in pediatric patients receiving chemotherapy over two sequential cycles.

SECONDARY OUTCOMES:
Chang is Safety from baseline | Up to 7 days
  Safety: based on medical review of adverse event reports and the results of vital sign measurements, electrocardiograms (ECGs)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Children's Hospital Colorado, Center for Cancer and Blood Disorders, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of South Florida, Tampa, Florida
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - UTSW/Childrens Medical Center, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Madigan Army Medical Center, Tacoma, Washington